CLINICAL TRIAL: NCT07340606
Title: The Role of Wolters Pulpitis Classification, Apical Periodontitis, and Artificial Intelligence-Assisted Diagnosis in Predicting the Success of Full Pulpotomy in Symptomatic Permanent Mature Molars: A Randomized Controlled Trial
Brief Title: The Role of the Pre-operative Condition and Artificial Intelligence-Assisted Diagnosis in Predicting the Success of Full Pulpotomy in Symptomatic Permanent Mature Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Mayand Amer Mohamed Yehia Amer, Principal Investigator, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIU-IRB-2425-036
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulpitis - Irreversible
Keywords: irreversible pulpitis; full pulpotomy; artificial intelligence; apical periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root Canal Treatment (Active Comparator): The patients allocated to this arm will receive conventional root canal treatment. They will be followed up for 1, 3, and 6 months to assess clinical and radiographic success.
  Interventions: Procedure: Conventional root canal treatment
- Full Pulpotomy (Experimental): The patients allocated to this arm will receive full pulpotomy. They will be followed up for 1, 3, and 6 months to assess clinical and radiographic success.
  Interventions: Procedure: Full pulpotomy

INTERVENTIONS:
Procedure: Conventional root canal treatment — The patients will receive conventional root canal treatment, which is the gold standard treatment protocol in cases with irreversible pulpitis.
  Arms: Root Canal Treatment
Procedure: Full pulpotomy — The patients will receive full pulpotomy as follows:
  -Under rubber dam isolation, the operator will perform caries removal, complete the access cavity preparation, achieve hemostasis in all canals, and apply the bioceramic material. The operator will seal the cavity with a glass ionomer restoration.
  Arms: Full Pulpotomy

SUMMARY:
This study aims to evaluate the effect of prognostic factors, such as the severity of pulpal inflammation, carious pulp exposure, and the presence of apical periodontitis, on the success of full pulpotomy in mature permanent molars with irreversible pulpitis. It also aims to investigate the role of artificial intelligence-assisted diagnosis in predicting the prognosis of full pulpotomy.

DETAILED DESCRIPTION:
* Patients with mature, permanent molars diagnosed with irreversible pulpitis will be enrolled in the study.
* The pre-operative pulpal status will be assessed using the American Association of Endodontists (AAE) classification and Wolters classification.
* Pre-operative digital radiographs will be taken, and radiographic caries depth will be assessed.
* The presence of pre-operative apical periodontitis will be recorded.
* An artificial intelligence software will process the pre-operative X-rays to assess the presence of carious pulp exposure and apical periodontitis.
* The patients will be randomly allocated to receive either full pulpotomy or conventional root canal treatment.
* The cases will be followed up for 1, 3, and 6 months to assess clinical and radiographic success. The accuracy of the AI software will be compared to the clinical findings of pulpal exposure after caries removal.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent molars with irreversible pulpitis.
* Presence of bleeding from all canals.
* The tooth is not periodontally compromised.

Exclusion Criteria:

* Non-vital teeth.
* Uncontrolled bleeding from any of the canals after ten minutes of application of hemostatic agent.
* Molars with immature roots.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Successful Cases | After 1, 3, and 6 months.
  * It will be measured as a percentage.
  * It will be decided according to the clinical and radiographic criteria of success and failure.
Diagnostic Accuracy (Sensitivity and Specificity) of an artificial intelligence software in detecting carious pulp exposure | On the day of the procedure
  The artificial intelligence (AI) software will process pre-operative radiographs to predict the presence of carious pulp exposure. The AI findings will be compared to the clinical findings of carious pulp exposure after caries removal. (Clinical findings of carious pulp exposure will be used as the gold standard).
  -The outcome will be reported as sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Ghobashy, Prof. Dr., Study Director — Misr International University; Mayand A Amer, B.D.S., Principal Investigator — Misr International University; Marwan S Ibrahim, B.D.S., Principal Investigator — Misr International University
Locations (2):
- Egypt (2):
  - Misr International University (MIU), Cairo
  - Misr International University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP